CLINICAL TRIAL: NCT04405583
Title: A Multicentre, International, Follow-up Study to Monitor the Efficacy and Safety of the Occlutech Atrial Flow Regulator in Heart Failure Patients
Brief Title: The AFteR Registry - Follow-up Study to Monitor the Efficacy and Safety of the Occlutech AFR in Heart Failure Patients
Acronym: AFR Registry
Status: Recruiting | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2020_01
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Occlutech AFR; Atrial Flow Regulator; Interatrial shunt device; Heart failure; HFrEF; HFpEF; Left-to-right shunt; Balloon atrial septostomy; MACNE; Device embolization; AFR; AFR Registry
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Occlutech Atrial Flow Regulator — The Occlutech Atrial Flow Regulator is an interatrial shunt device for transcatheter delivery.
  Other Names: Occlutech AFR

SUMMARY:
This study aims to monitor the safety and efficacy of Occlutech AFR device in patients with Heart Failure.

DETAILED DESCRIPTION:
This is a prospective, multicentre, international, follow-up registry to monitor the safety and the performance of the Occlutech AFR device in patients with Heart Failure, to identify unknown side effects and to assess the indications and contraindications for an AFR treatment. Efficacy and safety of implanted device(s) will be evaluated by vital signs, laboratory test, quality of life questionnaire, ECG, and echocardiography data over a follow-up period of 36 month after implantation.

Patients will be treated according to the instruction-for-use of the device and according to clinical routine. Procedures will be performed at sites having appropriate laboratory support and adequately trained imaging personnel. Procedures will be performed by physicians with experience in a wide range of interventional cardiology and structural heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent
2. Age ≥18 years
3. Presence of chronic symptomatic HF (NYHA class ≥ 2)
4. Left Atrial Pressure (LAP) > Right Atrial Pressure (RAP); with a gradient equal or more than 5 mmHg*
5. LVEF ≥ 15%. If LVEF is >40% (HFpEF), BMI corrected** NT-pro-BNP must be elevated ≥ 125 pg/mL. (BNP >35 pg/mL) or ≥ 365pg/ml (BNP > 105 pg/mL) for patients with atrial fibrillation (AF)
6. Stable guideline directed treatment according to latest applicable ESC guidelines for respective HF phenotypes for at least 1 months prior to informed consent

Exclusion Criteria:

1. Life expectancy < 1 year, or advanced heart failure defined as ACC/AHA Stage D heart failure, or listed for heart transplantation at time of baseline visit
2. Evidence of right heart failure defined (by ECHO) as:

   1. Severe Right Ventricular Dysfunction (TAPSE < 14 mm)
   2. Severe Right Ventricular Dilatation (RV volume ≥ LV volume)
   3. Severe pulmonary hypertension (PASP > 60 mm Hg)
3. Echocardiographic evidence of intra-cardia mass, thrombus or vegetation
4. Uncontrolled hypertension, Systolic Blood Pressure of >160 mmHg or Diastolic Blood Pressure ≥ 100mmHg, despite medical therapy at the time of screening visit.
5. Uncontrolled atrial fibrillation with resting heart rate >110bpm, despite medical therapy
6. Documented history of specific cardiomyopathy (obstructive hypertrophic, restrictive, infiltrative) or pericardial disease
7. Congenital heart defect that interferes with placement of the device, at the discretion of the Investigator.
8. Previous interventional or surgical atrial septal defect (ASD) or patent foramen ovale (PFO) closure interfering with the placement of the device
9. Current atrial septal defect, or anatomical anomaly (including > 10 mm atrial septal thickness or atrial septal aneurysm) on ECHO that precludes implantation of the device across the fossa ovalis (FO) of the interatrial septum
10. Clinically significant valvular heart disease:

    1. regurgitation grade ≥3+ or
    2. severe stenosis of mitral or tricuspid valves, or
    3. significant stenosis of aortic valves
11. Prior diagnosis of primary pulmonary hypertension
12. Severe Chronic Obstructive Pulmonary Disease (COPD) requiring oral steroid therapy or oxygen administration
13. History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within 6 months, or any prior stroke with persistent neurologic deficit, or any prior intracranial bleed, or known intracerebral aneurysm, AV malformation or other intracranial pathology increasing the risk of bleeding
14. Myocardial Infarction (MI) and/or coronary heart disease with indication for a coronary intervention or Coronary Artery Bypass Grafting (CABG) or within 2 months prior to informed consent.
15. ICD or right sided pacemaker placement within 2 months
16. Clinically significant coagulation disorder, at discretion of investigator
17. Patients with sepsis (local or generalized) or other acute infection(s) requiring systemic antibiotics in the two months prior enrollment
18. Chronic kidney disease currently requiring dialysis
19. Allergy to nickel and/or titanium and/or nickel/titanium-based materials, if not medically manageable
20. Allergy to anti-platelet, anti-coagulant or anti-thrombotic therapy
21. Participating in another investigational clinical trial that could interfere with this study, at the discretion of the investigator
22. Other clinically significant co-morbidities that make the patient unsuitable for study participation, at the discretion of the investigator

Note: * LA pressure is substituted by PCW at the right heart catheterization measure while patient is awaken

**"Corrected" refers to a 4% reduction in the NT-proBNP cutoff for every increase of 1kg/m2 in body mass index (BMI) above a reference BMI of 20kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 Heart Failure patients with reduced ejection fraction (HFrEF) or preserved ejection fraction (HFpEF), age ≥18 years, who gave their signed and dated informed consent will be included in the study analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects with at least one Major Adverse Cardiovascular and Neurologic Events (MACNE) in the 1 year following implantation. | 1 year
  MACNE includes all-cause mortality, stroke, systemic thromboembolism, open cardiac surgery or major endovascular repair, and major bleeding (BARC 3-5).

SECONDARY OUTCOMES:
Rate of subjects with at least one SAE/ (S)ADE at 12 months, 24 months and 36 months after implantation. | 3 years
Cardiovascular Events at 12 months, 24 months and 36 months after implantation. | 3 years
  Heart Failure hospitalization rate; Cardiovascular mortality; Unplanned HF admission or treatment intensification.
Device performance at 12 months, 24 months and 36 months after implantation. | 3 years
  Device placed in situ as assessed by the investigator; Patency: evidence of LEFT TO RIGHT shunt through the AFR device; Implant embolization and clinically significant device migration.
NYHA class status in comparison to Baseline. | 3 years
Subject QoL assessment using the KCCQ in comparison to Baseline. | 3 years
6 Minute Walk Test distance [m] in comparison to Baseline. | 3 years
Heart rhythm in comparison to Baseline | 3 years
Left Ventricular (LV), Right Ventricular (RV) and Left Atrial (LA) structure and function including strain derived indices in comparison to Baseline. | 3 years
Left Ventricular Ejection Fraction (LVEF) in comparison to Baseline. | 3 years
Tricuspid Annular Plane Systolic Excursion (TAPSE) in comparison to Baseline. | 3 years
Laboratory variables | 3 years
  Laboratory variables, including changes from baseline in: eGRF, NT-Pro-BNP [pg/ml]
Changes in heart failure related medication | 3 years
  reduction/increase of daily dose [%]
Relationship between pacemaker therapy and intra atrial shunt therapy | 3 years

CONTACTS AND LOCATIONS:
Locations (36):
- France (5):
  - CHU Besançon, Besançon
  - CHU Bourdeaux, Bourdeaux
  - CHU Lyon, Lyon
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Universitaire Rangueil, Toulouse
- Germany (10):
  - Knappschaftskrankenhaus Bottrop GmbH, Bottrop
  - Clinic Coburg, Coburg
  - University Clinic, Cologne
  - Helios Clinic Erfurt, Erfurt
  - Cardiologicum Hamburg, Hamburg
  - WKK Heide, Heide
  - University Clinic Jena, Jena
  - Hospital Osnabrueck, Osnabrück
  - Elbe Clinic Stade, Stade
  - University Clinic Tübingen, Tübingen
- Greece (5):
  - Hippokration Hospital Athens, Athens
  - Mitera Hospital Athens, Athens
  - Onassis Cardiac Surgery Center, Athens
  - European Interbalkan Medical Center, Thessaloniki
  - Hippokration Hospital of Thessaloniki, Thessaloniki
- Italy (2):
  - Careggi University Hospital, Florence
  - Centro Cardiologico Monzino, Milan
- Portugal (2):
  - Hospital de Santa Cruz, Carnaxide
  - Hospital de Santa Marta, Lisbon
- Dedinje Cardiovascular Institute, Dedinje, Serbia
- Tunisia (2):
  - Rabta Hospital, Tunis
  - The Military Hospital of Tunis, Tunis
- Turkey (Türkiye) (9):
  - Ankara Etlik Şehir Hastanesi, Ankara
  - Güven Hospital, Ankara
  - Hacettepe Üniversitesi Tip Fakültesi, Ankara
  - Firat University Hospital, Elâzığ
  - Binali Yildirim University Mengücek Gazi Training and Resear, Erzincan
  - Bezmialem Uni. Hospital, Fatih
  - İzmir City Hospital, Izmir
  - Kocaeli Üniversitesi Araştirma Ve Uygulama Hastanesi, Kocaeli
  - Namik Kemal University Hospital, Tekirdağ